CLINICAL TRIAL: NCT05842226
Title: THE EFFECT OF SYMPTOM MANAGEMENT EDUCATION GIVEN WITH MICRO TEACHING METHOD ENRICHED WITH STANDARD PATIENT IN PALLIATIVE CARE ON NURSING STUDENTS' KNOWLEDGE LEVEL, REFLECTIVE THINKING LEVEL AND THERAPEUTIC COMMUNICATION SKILLS
Brief Title: SYMPTOM MANAGEMENT EDUCATION GIVEN WITH MICRO TEACHING METHOD ENRICHED WITH STANDARD PATIENT IN PALLIATIVE CARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-06
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Palliative Care
Keywords: palliative care; micro teaching; standard patient; symptom management; nursing students

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Micro-teaching enriched with standard patient will be applied.
  Interventions: Other: Micro-teaching enriched with standard patient
- Control group (No Intervention): The control group will receive palliative care brochure for patients and their relatives.

INTERVENTIONS:
Other: Micro-teaching enriched with standard patient — The practice group will be shared the 4 most common symptoms in palliative care nursing: pain, fatigue, respiratory distress and loss of appetite. The practice group will be 5 groups and there will be 4 students in each group. During the practice, each student will provide patient education about only one symptom. The standard patient will participate in the intervention in the application laboratory and the students will participate in the intervention in the computer environment. Video recordings will be taken while the students are giving education. After watching the experts, peers and their own video with the micro-teaching group evaluation form, the student himself/herself will make an evaluation. At the same time, a lecturer from outside the research will fill in the Standard Patient Check-List Evaluation Form. The application will be repeated one week later.
  Arms: Intervention group

SUMMARY:
The study was planned as a randomized controlled pre-test, post-test intervention study to determine the effect of symptom management training in palliative care given with micro-teaching method enriched with standard patient on nursing students' knowledge levels, reflective thinking levels and therapeutic communication skills related to palliative care.

DETAILED DESCRIPTION:
Sample of study was calculated as 36 using G*Power Software (ver. 3.1.9.2) for 80% power and medium effect size (f=0.40) at 95% confidence level in line with the data of Lin et al. The experimental and control groups were planned as 20 students each with a 10 percent loss. Participants were assigned to the experimental and control groups by the stratified randomization method. The locks were assigned to layers using Microsoft Excel. A pre-test will be applied to both groups. The control group will receive palliative care brochure for patients and their relatives.The practice group will be shared the 4 most common symptoms in palliative care nursing: pain, fatigue, respiratory distress and loss of appetite. The practice group will be 5 groups and there will be 4 students in each group. During the practice, each student will provide patient education about only one symptom. The standard patient will participate in the intervention in the application laboratory and the students will participate in the intervention in the computer environment. Video recordings will be taken while the students are giving education. After watching the experts, peers and their own video with the micro-teaching group evaluation form, the student himself/herself will make an evaluation. At the same time, a lecturer from outside the research will fill in the Standard Patient Check-List Evaluation Form. The application will be repeated one week later. After all the applications, the students will watch the video of their own 2 more times and the post-test will be applied to both groups. After one month, a retention test will be applied to the students in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Students taking palliative care course for the first time,
* Students who agreed to participate in the study,

Exclusion Criteria:

* Students who have already taken the palliative care course,
* Students who answered the data collection forms incompletely,
* Students who do not want to continue the research,
* Students who missed even one of the theoretical or practical sessions of the study.
* Students with experience of caring for a palliative care patient

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
KNOWLEDGE LEVEL | 2 months
  A knowledge test on symptom management and communication in palliative care was developed by the researcher. It consists of 25 questions.
REFLECTIVE THINKING LEVEL | 2 months
  Scale for Determining the Level of Reflective Thinking will be used. It is a 16-item 5-point Likert-type scale consisting of four sub-dimensions. Its sub-dimensions are habituation, comprehension, reflection and critical reflection.
THERAPEUTIC COMMUNICATION SKILLS | 2 months
  Therapeutic Communication Skills Scale for Nursing Students will be used. It is a 7-point Likert scale consisting of a total of 16 items, including 7 items in the NonTherapeutic Communication Skills sub-dimension, 6 items in the Therapeutic Communication Skills 1 sub-dimension, and 3 items in the Therapeutic Communication Skills 2 sub-dimension.

SECONDARY OUTCOMES:
Micro Teaching Group Evaluation Form | 2 weeks
  It was created by the researcher. It will be used for self-assessment by experts, peers and the student during the implementation.
Standard Patient Evaluation Form | 2 weeks
  Created by the researcher. It will be filled in by specialists during standardized patient practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Tayaz, Ankara, Mamak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No